CLINICAL TRIAL: NCT01783860
Title: Study of the Effect of Oral Azithromycin on Posterior Blepharitis
Brief Title: Oral Azithromycin Versus Doxycycline in Posterior Blepharitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90-01-124-13076
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-12

CONDITIONS: Posterior Blepharitis
Keywords: Azithromycin; Doxycycline; Posterior Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Azithromycin (Experimental): Two 250 mg capsules (500 mg) of Azithromycin for the first day and 250mg/day for the next 4 days.
  Interventions: Drug: Azithromycin
- Doxycycline (Active Comparator): Oral doxycycline 100mg capsule every 12 hours for one month
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Azithromycin
  Other Names: Azithromycin (Razak Co., Tehran)
  Arms: Oral Azithromycin
Drug: Doxycycline
  Other Names: Doxycycline (Kimidarou Co., Tehran)
  Arms: Doxycycline

SUMMARY:
One hundred patients with the diagnosis of posterior blepharitis based on history taking and proper physical examinations by two experienced ophthalmologists will include in the study.

Patients will diagnose with posterior blepharitis if they score at least one in two symptoms (based on a subjective grading scale) and two signs (based on an objective grading scale) of posterior blepharitis according to study criteria. Patients will exclude if they have the following criteria: age< 12 years old,history of previous ocular or lacrimal surgery,previous usage of contact lenses,any history of ocular allergy,history of systemic diseases with ocular involvement (except rosacea), history of usage of topical or systemic antibiotic in the last month, pregnancy or lactating mothers, liver failure and any history of sensitivity to cyclines.

Qualified patients then randomly receive oral azithromycin (2 of 250 mg capsules for the first day and 250mg for the next 4 days) or oral doxycycline (100mg capsule every 12 hours for one month) in a double-blinded fashion. each patients in both treatment groups will accurately instruct to apply warm compress and eyelid scrubbing 2 times a day for 5 minutes each in the treatment period. Symptoms and signs were recorded for each patient in two treatment groups at baseline visit (before treatment) and then in the days 7, 31, 37 and 61 after treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients were diagnosed with posterior blepharitis if they scored at least one in two symptoms (based on a subjective grading scale) and two signs (based on an objective grading scale) of posterior blepharitis according to study criteria

Exclusion Criteria:

Patients were excluded if they had the following criteria: age< 12 years old,history of previous ocular or lacrimal surgery,previous usage of contact lenses,any history of ocular allergy,history of systemic diseases with ocular involvement (except rosacea), history of usage of topical or systemic antibiotic in the last month, pregnancy or lactating mothers, liver failure and any history of sensitivity to cyclines

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Study Director — Tehran University of Medical Sciences
Locations (1):
- Rassoul Akram Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Kashkouli MB, Fazel AJ, Kiavash V, Nojomi M, Ghiasian L. Oral azithromycin versus doxycycline in meibomian gland dysfunction: a randomised double-masked open-label clinical trial. Br J Ophthalmol. 2015 Feb;99(2):199-204. doi: 10.1136/bjophthalmol-2014-305410. Epub 2014 Aug 19. PMID 25138765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 100 patients were selected from the eye clinic of Rasoule-Akram hospital during the study period. The patients were recruited sequentially.
Pre-assignment Details: Patients were excluded if they had: age< 12 years,history of ocular or lacrimal surgery,previous usage of contact lenses,history of ocular allergy or systemic diseases with ocular involvement, history of usage of topical or systemic antibiotic in the last month, pregnant or lactating mothers, liver failure and history of sensitivity to Cyclines.
Groups:
- Doxycycline: Oral doxycycline 100mg capsule every 12 hours for one month
  Doxycycline :
- Oral Azithromycin: Two 250 mg capsules (500 mg) of Azithromycin for the first day and 250mg/day for the next 4 days.
  Azithromycin :
Period: Overall Study
Arm/Group | Doxycycline | Oral Azithromycin
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Oral Azithromycin | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 46 | 43 | 89
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change of Blepharitis Symptoms Score
Description: Five main ocular symptoms of posterior blepharitis (itching, foreign body sensation, dryness, burning, and lid swelling) will be asked of each patient and graded at baseline, and days 7, 31, 37 and 61 after treatment. For each item there was a question with scale from zero to three (zero for no symptom three for maximum symptom). Therefore, maximum score for symptoms was 15 (worse outcome) and minimum score for symptoms was zero (better outcome). Finally, we reported a change in total score calculated as the latest time point (61 days) minus the earliest time point.
Time Frame: Change from the baseline until 61 days after treatment
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
score | 1.8 (2.5) | 2.8 (2.2)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p = 0.03, t-test, 1 sided

2. Secondary Outcome: Main Ocular Signs
Description: lid margin debris, lid margin redness, Meibomian gland (MG) secretion, occluded MG, conjunctival redness, tear brake up time and ocular surface staining at Baseline, and days 7, 31, 37 and 61 after treatment were measured. For each items there was a question with scale form zero to three (zero for no sign to three for maximum sign). Therefore, maximum score for signs was 21 (worse outcome) and minimum score was zero (better outcome). We calculated a total score for signs. Finally, we reported a change in total score calculated as the latest time point (61 days) minus earliest time point.
Time Frame: Change from baseline until 61 days after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
units on a scale | 4.7 (2.3) | 5.7 (2.0)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p = 0.01, t-test, 1 sided

3. Primary Outcome: Change of Symptoms and Signs Scores (Difference Between Total Score of First Time and 61 Days Later), Total Severity Score
Description: Total severity score was a combined score of symptoms and signs. For symptoms, there were five items and for signs there were seven items. Each items had three scales form Zero (no symptom) to three (severe symptom). Therefore, there was 12 items to calculate total severity score. Maximum score was 36 (worse outcome) and minimum score was zero (better outcome). A change in total severity score calculated as the latest time period (61 days) minus earliest time point.
Time Frame: zero time and 61 days later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
units on a scale | 6.5 (4.1) | 8.6 (3.6)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p = 0.007, t-test, 1 sided

4. Other Pre Specified Outcome: Change of Total Severity Score Between Baseline and 7 Days Later
Description: Total severity score was a combined score of symptoms and signs. For symptoms, there were five items and for signs there were seven items. Each items had three scales form Zero (no symptom) to three (severe symptom). Therefore, there was 12 items to calculate total severity score. Maximum score was 36 (worse outcome) and minimum score was zero (better outcome). A change in total severity score calculated as the latest time period (7 days) minus earliest time point.
Time Frame: baseline and 7 days later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
units on a scale | 3.9 (2.5) | 4.3 (2.6)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

5. Other Pre Specified Outcome: Change of Total Severity Score Between Baseline and 31 Days Later
Description: Total severity score was a combined score of symptoms and signs. For symptoms, there were five items and for signs there were seven items. Each items had three scales form Zero (no symptom) to three (severe symptom). Therefore, there was 12 items to calculate total severity score. Maximum score was 36 (worse outcome) and minimum score was zero (better outcome). A change in total severity score calculated as the latest time period (31 days) minus earliest time point.
Time Frame: baseline and 31 days later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
units on a scale | 5.2 (2.4) | 6.4 (2.6)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p = 0.02, t-test, 1 sided

6. Other Pre Specified Outcome: Change of Total Severity Score Between Baseline and 37 Days Later
Description: Total severity score was a combined score of symptoms and signs. For symptoms, there were five items and for signs there were seven items. Each items had three scales form Zero (no symptom) to three (severe symptom). Therefore, there was 12 items to calculate total severity score. Maximum score was 36 (worse outcome) and minimum score was zero (better outcome). A change in total severity score calculated as the latest time period (37 days) minus earliest time point.
Time Frame: baseline and 37 days later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Oral Azithromycin
Number analyzed (Participants) | 50 | 50
units on a scale | 6.3 (3.2) | 7.4 (3)
Statistical Analysis 1: Comparison: Doxycycline vs Oral Azithromycin; Test type: Superiority or Other; p = 0.08, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Doxycycline | Oral Azithromycin
Serious Adverse Events (participants affected / at risk) | 12/50 | 3/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxycycline (N=50) | Oral Azithromycin (N=50)
vomiting and loss of appetide (Gastrointestinal disorders) | 12 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes